CLINICAL TRIAL: NCT01587001
Title: The Effect of an Oral Antioxidant, N-Acetyl-L-Cysteine, on Inflammatory and Oxidative Stress Markers in Pulmonary Sarcoidosis
Brief Title: The Effect of N-Acetyl-L-Cysteine, on Inflammatory and Oxidative Stress Markers in Pulmonary Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22219201
Record Dates: First submitted 2012-01-10; First posted 2012-04-27 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Sarcoidosis; oxidative stress; anti-oxidant
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral N-acetyl-cysteine (Active Comparator): oral NAC 900mg three times daily for 8 weeks
  Interventions: Dietary Supplement: N-acetyl-cysteine
- Matching Placebo (Placebo Comparator): oral placebo three times daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: N-acetyl-cysteine — 900mg three times daily for 8 weeks
  Arms: Oral N-acetyl-cysteine
Drug: Placebo — Matching placebo three times daily for 8 weeks.
  Arms: Matching Placebo

SUMMARY:
This is a pilot study investigating the effect of an antioxidant, N-Acetyl-L-Cysteine (NAC), on inflammation and oxidative stress in sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a granulomatous lung disease predominantly affecting the lungs. Reactive oxidative species are produced secondary to oxidative stress and inflammation and can affect key cellular processes. The investigators have shown a role for oxidative stress in chronic beryllium disease (CBD), a granulomatous disease that resembles sarcoidosis, and have also shown that antioxidant therapy reduces inflammation in CBD. Oxidative stress also plays a role in sarcoidosis but the exact mechanism and potential effect of antioxidant therapy on sarcoidosis is unknown. The investigators propose conducting a pilot study investigating the effect of an antioxidant, N-Acetyl-L-Cysteine (NAC), on inflammation and oxidative stress in sarcoidosis. The investigators will measure and compare markers of inflammation and oxidative stress in the lungs of sarcoidosis patients before and after treatment with NAC. The results of this study will prepare the investigators for a larger study investigating the role of NAC as a therapy for sarcoidosis with changes in lung function and x-ray as our primary outcome. This will provide the investigators with a new non-toxic therapy for sarcoidosis that can be used on its own or to supplement other therapies minimizing their toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven sarcoidosis.
* Pulmonary parenchymal involvement with a Scadding chest x-ray stage II, III or IV.
* Abnormal spirometry and/or DLCO (< 80% of predicted).
* Consenting adults : Age 18 years and above

Exclusion Criteria:

* Positive lung washing or biopsy cultures for fungi or mycobacterial disease;
* Presence of other co-morbid conditions that may affect the patient's outcome.
* Patient inability to undergo venipuncture and BAL procedures.
* Current use of tobacco (smoking or otherwise) in the past 6 months
* Treatment with immunosuppressive therapy within the past 6 months.
* On oral anti-oxidant supplements.
* Active peptic ulcer disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Hamzeh, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral N-acetyl-cysteine | Matching Placebo
Started | 14 | 3
Completed | 8 | 2
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Insufficient samples to complete testing | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral N-acetyl-cysteine | Matching Placebo | Total
Number analyzed (Participants) | 11 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9) | 52 (13) | 53 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 11 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 11 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Bronchoalveolar Lavage (BAL) and Peripheral Blood Mononuclear Cells (PBMC) TNF-α Levels
Description: Baseline peripheral blood mononuclear cells and bronchoalveolar lavage (BAL) lymphocyte percentages and lipopolysaccharide (LPS) stimulated tumor necrosis factor-α levels (pg/ml)
Time Frame: 8 weeks of anti-oxidant therapy
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oral N-acetyl-cysteine | Matching Placebo
Number analyzed (Participants) | 8 | 2
pg/ml
  Mean baseline BAL cell TNF-a | 40767 (25684) | 39938 (12033)
  Mean follow-up BAL cell TNF-a | 45176 (17910) | 25671 (12203)
  Mean baseline PBMC cell TNF-a | 2775 (2292) | 637 (404)
  Mean follow-up PBMC cell TNF-a | 3387 (2481) | 969 (135)

2. Secondary Outcome: Bronchoalveolar Lavage (BAL) Cell Glutathione (GSH) Levels
Description: We measured changes at baseline and at 8 weeks in BAL whole cell total GSH levels and cellular 8-OHdG before and after treatment with NAC/placebo.
Time Frame: 8 weeks of anti-oxidant therapy
Measure: Mean (Standard Deviation); unit: nmol/mg protein
Arm/Group | Oral N-acetyl-cysteine | Matching Placebo
Number analyzed (Participants) | 8 | 2
nmol/mg protein
  Baseline visit | 5.93 (2.94) | 9.39 (2.06)
  8 week visit | 9.42 (3.64) | 4.28 (0.12)

ADVERSE EVENTS:
Arm/Group | Oral N-acetyl-cysteine | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 0/11 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No